CLINICAL TRIAL: NCT05320055
Title: Less Postoperative Pain and Length of Stay After Robotic-assisted Laparoscopic Transabdominal Repair With Retro Rectus Mesh Placement (rTARUP) Compared With Laparoscopic Intraperitoneal Onlay Mesh Repair (IPOM) for Small and Medium-sized Ventral Hernias
Brief Title: Pain and Readmission After Lap IPOM vs. Robotic Ventral Hernia Repair
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Mette Willaume, Staff specialist, MD, PhD, Bispebjerg Hospital
Other Study IDs: IPOM vs TARUP
Record Dates: First submitted 2022-04-01; First posted 2022-04-11 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Hernia, Ventral
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IPOM: receiving laparoscopic intraperitoneal onlay mesh repair
  Interventions: Procedure: robotic repair
- rTARUP: recieving robotic assited retromuscular repair
  Interventions: Procedure: robotic repair

INTERVENTIONS:
Procedure: robotic repair — robotic assisted retromuscular hernia repair

SUMMARY:
Comparison of results after rTARUP and lap IPOM in patients with small- and medium-sized ventral hernia. Retrospective cohort study of consecutive patients undergoing rTARUP or IPOM repair for small or medium-sized primary ventral and incisional hernias. The primary outcome was the postoperative need for transverse abdominis plane (TAP) block or epidural catheter, secondary outcomes were 30-day complications, and length of stay. All patients underwent elective surgery and were followed for 30 days postoperatively.

DETAILED DESCRIPTION:
Single-center retrospective cohort study of consecutive patients undergoing rTARUP or IPOM repair for small or medium-sized primary ventral and incisional hernias. The primary outcome was the postoperative need for transverse abdominis plane (TAP) block or epidural catheter, secondary outcomes were 30-day complications, and length of stay. All patients underwent elective surgery and were followed for 30 days postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing elective minimally invasive repair for small or medium-sized primary ventral or incisional hernia repairs at one academic hernia center with an unrestricted patient referral.

Consecutive patients undergoing IPOM (December 1st, 2017 - December 1st, 2018) and rTARUPrRetrorectus (March 1st, 2021 - June 1st, 2021).

Exclusion Criteria:

* open repairs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population is all patients referred from primary sector and eligible for laparoscopic primary ventral or incisional hernia repair
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
epidural blockade or TAP block | 0-1 postoperative day
  postoperative pain requiring epidural or TAP block

SECONDARY OUTCOMES:
readmissison | 30 days
  if the patients get readmitted during the follow-up
complications | 30 days
  if the patients get any medical or surgical complication during the follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Mette Willaume, phd, Principal Investigator — University of Copenhagen, Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Christoffersen MW, Jorgensen LN, Jensen KK. Less postoperative pain and shorter length of stay after robot-assisted retrorectus hernia repair (rRetrorectus) compared with laparoscopic intraperitoneal onlay mesh repair (IPOM) for small or medium-sized ventral hernias. Surg Endosc. 2023 Feb;37(2):1053-1059. doi: 10.1007/s00464-022-09608-w. Epub 2022 Sep 15. PMID 36109358